CLINICAL TRIAL: NCT00604838
Title: Pivotal Study of the Al-ASense Study Protocol
Brief Title: Pivotal Study of the Al-Sense Study Protocol
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Clinical studies manager, Common Sense Ltd.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AlSense-Pivot101
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Last update posted 2008-01-30 (Estimated); Status verified 2008-01

CONDITIONS: Amniotic Fluid Leakage
Keywords: amniotic fluid leakage; urinary incontinence; pregnancy; home test; vaginal wetness
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- I (Experimental)
  Interventions: Device: AL-SENSE Diagnostic Absorbent Panty liner

INTERVENTIONS:
Device: AL-SENSE Diagnostic Absorbent Panty liner — worn for 12 hours
  Other Names: AL-SENSE Amniotic Leak Test Kit
Device: AL-SENSE Diagnostic Absorbent Panty liner — Diagnostic Absorbent Panty liner (AL-SENSE Amniotic Leak Test Kit), developed by Common Sense Ltd worn for 12 hours

SUMMARY:
The purpose of this study is to demonstrate that the Diagnostic Absorbent Panty liner (AL-SENSE Amniotic Leak Test Kit), developed by Common Sense Ltd., can distinguish between wetness sensed by pregnant women that is caused by amniotic fluid leakage and that which is caused by urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 45 years.
* minimum 16 weeks of pregnancy.
* willing to sign the informed consent form.
* arrived at the obstetric department reporting a feeling of vaginal wetness (undetermined whether this is amniotic fluid leakage or urinary incontinence).

Exclusion Criteria:

* experienced intermittent vaginal bleeding between the 2nd and 3rd trimester.
* have had sexual relations within the last 12 hours.
* unable or unwilling to cooperate with study procedures.
* used the AL-SENSE before joining this study.
* diagnosed with Bacterial Vaginosis or Trichomonas infection within the last 3 days.
* uses vaginal products such as some douching formulas, some antibiotic treatments which reduce lactobacillus population.
* uses drugs which reduce estrogen level such as tamoxifen or drugs that dry out the mucous membranes, such as antihistamines
* on a diet of alkalizing foods such as Alkalive™ Green, which may cause elevation of the vaginal pH level.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 330 (Actual)
Dates: Start 2006-05; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
presence or absence of a blue-green stain on a yellow background as yielded by the AL-SENSE and observed by the patient. | up to 12 hours

SECONDARY OUTCOMES:
presence or absence of a blue-green stain on a yellow background as yielded by the AL-SENSE and observed by the clinician and a measurement of patient comfort while using AL-SENSE and reading the results. | up to 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Bornstein, MD, Principal Investigator — Western Galilee Hospital-Nahariya; Yoram Sorokin, MD, Principal Investigator — Wayne State University / Hutzel Women's Hospital
Locations (2):
- Wayne State University / Hutzel Women's Hospital, Detroit, Michigan, United States
- Western Galilee Hospital-Nahariya, Nahariya, Israel

REFERENCES:
- [Background] Watanabe T, Minakami H, Itoi H, Sato I, Sakata Y, Tamada T. Evaluation of latex agglutination test for alpha-fetoprotein in diagnosing rupture of fetal membranes. Gynecol Obstet Invest. 1995;39(1):15-8. doi: 10.1159/000292368. PMID 7534254
- [Background] Garite TJ, Gocke SE. Diagnosis of preterm rupture of membranes: is testing for alpha-fetoprotein better than ferning or nitrazine? Am J Perinatol. 1990 Jul;7(3):276-8. doi: 10.1055/s-2007-999500. PMID 1695510
- [Background] Kishida T, Yamada H, Negishi H, Sagawa T, Makinoda S, Fujimoto S. Diagnosis of preterm premature rupture of the membranes using a newly developed AFP monoclonal antibody test kit. Eur J Obstet Gynecol Reprod Biol. 1995 Jan;58(1):67-72. doi: 10.1016/0028-2243(94)01973-b. PMID 7538939
- [Background] Rochelson BL, Rodke G, White R, Bracero L, Baker DA. A rapid colorimetric AFP monoclonal antibody test for the diagnosis of preterm rupture of the membranes. Obstet Gynecol. 1987 Feb;69(2):163-6. PMID 2433650